CLINICAL TRIAL: NCT01158768
Title: Questionnaire to Study Impacts in the Health of the Woman in the Climateric's Phase, Victim of Domestic and/or Sexual Violence
Brief Title: Questionnaire to Study Violence Against Women in the Climateric's Phase.
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Núcleo de Estudos Sobre Violência e Humanização da Assistencia à Saúde (Other)
Responsible Party: Angela Maggio da Fonseca, University of Sao Paulo General Hospital
Other Study IDs: 180/09.1
Record Dates: First submitted 2010-05-14; First posted 2010-07-08 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2009-03

CONDITIONS: Comorbidity; Domestic Violence; Sexual Abuse
Keywords: domestic violence in childhood/adolescence; comorbidities; climactery; domestic violence against women; trauma questionnaire; Violence

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Violence, Comorbidity

SUMMARY:
Objectives - To construct and validate a questionnaire evaluating violence suffered by women during any phase of their lives and health repercussions during climactery.

Method: A controlled study with the application of a questionnaire at the Outpatient Clinics for Endocrine Gynecology and Climactery of the University Hospital (Hospital das Clínicas) of the Medicine College of the University of São Paulo (FMUSP), Brazil, performed during 2009 for 124 women aged between 40 and 65 years, who were victims of domestic and/or sexual violence, distributed in three groups regarding the phase in which their experience with violence occurred: 1. Violence exclusively during childhood/adolescence; 2. During adulthood; 3. Throughout all phases. The instrument encompasses 13 key questions and 21 sub items evaluating: 1. Place of residence and who the woman lives with; 2. Start, frequency and type of violence; 3. Search for health assistance and report of the violence; 4. Violence and number of affections; 5. Violence and Menopausal Kupermann Index (IMK).

Results: The instrument presented Cronbach Alpha=0.82, reliability among examiners (+0,80), and good possibility to be reproduced. Average age of the women was 55,8 years (±6,6), menopause at -45,4 years in average, in the control Group (GC) it was 48,1 years; first sexual intercourse 19,5 years (GC = 21,0); menarche 13,1 years, and average BMI (Body Mass Index) 28,5 (±2,8), similar to the GC, but frequent violence during adulthood showed a BMI of 30,0 (±2,8). Women who were submitted to violence exclusively: during childhood 14,5%; adolescence 1,6%; adulthood 41,9%, during all phases of their lives 42,0%. Women subjected to violence during childhood/adolescence (58,1%) presented an average of 5,1 affections; during adulthood, 4,6 and 4,4 for both phases. Sexual violence (43,5%) and other types of violence both present average affections (4,60) but represent a significative impairment of sexual life. There were significative associations between suffering any type of violence during all phases of their lives, sexual violence during any phase of their lives and a serious IMK. Among those women, 80,6% did not search health services due to the violence suffered.

Conclusion: The questionnaire presents good internal consistency and a validated construction, can be easily reproduced and is indicated to evaluate the consequences of domestic and/or sexual violence on women´s health during climactery.

DETAILED DESCRIPTION:
The score for each dominium varied from 0 to 100 and the higher the score the worst is past experience with mistreats. Scores for each dominium were then compared to groups of patients previously defined.We employed statistic tests for two independent samples (Mann-Whitney). For all the tests we fixed in 0,05 or 5% the level of rejection of the null hypothesis. In order to characterize the study sample, patients were defined according to characteristics including anthropometric, climacteric and lifestyle features. Quantitative variables were described according to the average and the respective patter deviation, median and minimum and maximum values. Qualitative variables were described by simple percentages.

Questionnaire designed to analyze "Impacts on Women's Health during the climactery phase if victim of domestic or sexual violence" by Moraes & Fonseca, 2009 This is a two part set. If the woman suffered violence during childhood and;or adolescence, she will answer the Portuguese version of Childhood Trauma Questionnaire, which is a self applied instrument for adolescents and adults investigating history of abuse and negligence during childhood and adolescence. The instrument was translated, adapted and validated the questionnaire contents for a Portuguese version with the original name of "Questionário Sobre Traumas na Infância" (Childhood Trauma Questionnaire) (annex 1), by Grassi-Oliveira R et al, 2006.

If the woman was subjected to violence during her life, especially during adulthood, she will answer the questionnaire on "Impacts on Women's Health during Climactery Phase, if victim of domestic or sexual violence", elaborated and validated by Moares &¨Fonseca, 2009.

ELIGIBILITY:
Inclusion Criteria:

* Women (during the ages of 40 to 65 years) who were or are victims of domestic and/or sexual violence

Exclusion Criteria:

* Women who were not victims of domestic and/or sexual violence.
* Women that were not 40 to 65 years.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women (during the ages of 40 to 65 years) who were or are victims of domestic and sexual violence seeking attention at the outpatient clinic for Endocrines Gynecology and Climactery - University of Sao Paulo General Hospital during 2009.
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Number of comorbidities present in the climacteric phase and intensity of symptoms in women victims of domestic violence | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Fonseca, Assoc Prof, Study Director — University of Sao Paulo General Hospital; Sandra Dircinha TA Moraes, Post-Doc, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Hospital das Clinicas of the Medicine College of the University of São Paulo, São Paulo, São Paulo, Brazil